CLINICAL TRIAL: NCT03134001
Title: Evaluation of Oral Patient-Controlled Analgesia (PCA) Device - PCoA™ Acute , for Hospitalized Patients With Post-operative Pain
Brief Title: Evaluation of Oral PCA Device - PCoA™ Acute
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dosentrx Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PCoAAcute001
Record Dates: First submitted 2017-04-25; First posted 2017-04-28 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-04

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Study includes 2 groups: test group comprised patients receiving oral analgesics via the PCoA™ Acute and control group of nurse providing analgesics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Patients receiving oral analgesics via the PCoA™ Acute device
  Interventions: Device: patients receiving oral analgesics via the PCoA™ Acute
- Control Group (No Intervention): Patients receiving oral analgesics by nurse, upon request

INTERVENTIONS:
Device: patients receiving oral analgesics via the PCoA™ Acute — PCoA™ Acute is an oral PCA device, designed to provide safe and easy-to-use pain medication at the bedside. It identifies patients by Radio Frequency Identification (RFID) technology and provides pill dispensing upon patient's request.
  Arms: Test Group

SUMMARY:
Randomized, open label, controlled pilot clinical study comprised hospitalized post operative patients receiving oral analgesics. The study aims to evaluate the safety, efficacy and usability of a novel pill dispensing system - PCoA™ Acute and compare it to the conventional procedure of nurse providing analgesics.

ELIGIBILITY:
Inclusion Criteria:

1. Operative procedure with at least 3 days' hospital stay.
2. Planned post-operative pain therapy with oral medication using a strong opioid.
3. No contra-indication for opioid therapy.
4. No contra-indication for oral pain therapy.
5. Patient was able to understand and complete the questionnaire.
6. Patient signed an informed consent form.

Exclusion Criteria:

1. Opioid or drug addiction. 2. Opioid intolerance. 3. Pain therapy using IV PCA or infusion. 4. Rejection of opioid therapy. 5. Not able to swallow medicine.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2015-11-30 (Actual)

PRIMARY OUTCOMES:
PCoA™ Acute safety | 48 hr
  No pill overdose, No pills malformation upon dispensing, No pill inhalation during pill sucking, 4. No adverse events
PCoA™ Acute efficacy | 48hr
  Success rate of 90% for pill intake upon patient's request, No critical device malfunction, Time of pill intake reduced by at least 50% in the test group compared to the control group
PCoA™ Acute usability | 48hr
  At least 80% of patients and medical staff are satisfied with device use and will recommend its use for their colleagues

SECONDARY OUTCOMES:
Number of pill intakes during the study | 48hr
  Number of pain medications obtained by the patients during the study

IPD SHARING:
Plan to Share IPD: Undecided